CLINICAL TRIAL: NCT04223206
Title: K2DTD75 - ALTIS "Alimento Funzionale a Base di Lens Culinaris Tipico Del Territorio Pugliese ed Innovativo Per la Salute" - Regione Puglia "INNONETWORK 2017"
Brief Title: Innovative Functional Food Based on Apulian Lens Culinaris for Contrasting Sarcopenia in Dialysis Patients
Acronym: ALTIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: University of Bari Aldo Moro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K2DTD75_ALTISnefro
Record Dates: First submitted 2019-12-17; First posted 2020-01-10 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2021-01

CONDITIONS: Hemodialysis; Sarcopenia
Keywords: uremic toxins; gut microbiota dysbiosis; sarcopenia; hemodialysis
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemodialysis with sarcopenia (Experimental): 10 HD patients, affected by sarcopenia will a undergo 3-months supplementation with NATURLENS
  Interventions: Dietary Supplement: NATURLENS
- Controls (No Intervention): 10 HD patients, affected by sarcopenia will be followed for 3 months without any supplementation

INTERVENTIONS:
Dietary Supplement: NATURLENS — Oral administration of dietary supplement (26 g/day) to dissolve in 100 or 150 mL of water
  Arms: Hemodialysis with sarcopenia

SUMMARY:
The objective of the pilot study is to validate the clinical use of a dietary supplement for contrasting sarcopenia in dialysis patients.

The study aims at evaluating the effects of a nutritional supplement, consisting of flour from Lens culinaris of Altamura IGP, pea proteins and vitamins (A, B12, D, E) by achieving the following objectives:

* Reduction of sarcopenia conditions, through improvement of nutritional and anthropometrical levels
* Decrease of the serum levels of microbiota-derived uremic toxins
* Reduction of intestinal permeability and inflammatory markers

ELIGIBILITY:
Inclusion Criteria:

* patients > 60 years old
* omnivore controlled normocaloric diet (30 Kcal/kg ideal weight)
* patients with chronic kidney disease (CKD) and routine hemodialysis or peritoneal dialysis
* patients with primary sarcopenia identified with score ≥ 4 at SARC-F Questionnaire
* informed consent signed

Exclusion Criteria:

* participation to another clinical trial
* limb removal by amputation
* altered blood sugar level (HbA1c>8.0%) or type I diabetes mellitus
* neoplastic events in the last 5 years
* gut, systemic or autoimmune chronic inflammatory pathologies
* use of antibiotics or probiotics up to 30 days prior to recruitment
* life expectancy of less than one year
* treatment with corticosteroids or immunosuppressive drugs (excluded prednisone at dose <5 mg at day)
* positivity to hepatitis B and C virus, HIV1/2 and syphilis
* oxygen saturation in the blood at rest <93%
* alcohol or drug abuse in the last 3 years
* clinically important alterations of the following laboratory parameters: hemoglobin <9.0 g / dL, white blood cells <2.500 / μl, platelet count <100.000 / μl, AST and ALT> 3 times the upper limit of the norm, coagulopathy (INR> 1.3 ) not due to a reversible cause (eg Warfarin and / or factor Xa inhibitors)
* uncontrolled hypertension (resting systolic blood pressure> 180 mmHg or diastolic blood pressure> 110 mmHg)
* unstable angina pectoris, severe peripheral artery disease, coronary bypass surgery, angioplasty or acute major cardiocirculatory diseases in the previous 3 months
* definite congestive heart failure class III or IV (NYHS) or ejection fraction <25%
* severe pulmonary dysfunction: acute exacerbation of chronic obstructive pulmonary disease in phase III or IV (Gold classification) and / or PaO2 levels <60 mmHg
* significant intestinal malabsorption due to partial ileal bypass or other causes
* score ≤ 24 at the Mini Mental State Examination (MMSE) or presence of cognitive or linguistic limits that prohibit informed consent or possible elements of study
* diagnosis of disabling neurological disorder, including Parkinson's disease, amyotrophic lateral sclerosis, multiple sclerosis, cerebrovascular accident with residual deficits (for example, muscle weakness or gait disorder), dementia or any psychiatric condition that reduces protocol compliance
* have a history or evidence of any condition, therapy, laboratory abnormality or other circumstances that could confuse the results of the study or interfere with the patient's participation throughout the duration of the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of muscle mass | 3 months
  Change of muscle mass by bioelectrical impedance assessment (BIA)

SECONDARY OUTCOMES:
Change of sarcopenia conditions | 3 months
  Change of sarcopenia assessed by the European Working Group on Sarcopenia in Older People (EWGSOP) guidelines through the SARC-F (Strength, Assistance with walking, Rise from a chair, Climb stairs and Falls) questionnaire. The SARC-F scale scores range from 0 to 10 (i.e. 0-2 points for each item; 0=best to 10=worst) and represents no sarcopenia (0-3) and sarcopenia (4-10).
Change of Mini Nutritional Assessment (MNA) score | 3 months
  Measurement of MNA questionnaire (12-14 points, normal nutritional status; 8-11 points, at risk of malnutrition; 0-7, malnourished)
Change of anthropometric parameter | 3 months
  Measurement of the arm circumference (cm)
Change of body mass index (BMI) | 3 months
  Measurement of BMI (kg/m^2)
Change of gastrointestinal symptoms | 3 months
  Change of gastrointestinal symptoms assessed by Gastrointestinal Symptom Rating Scale (GSRS) questionnaire (15 items scored 1-7 each, 1 representing the best and 7 the worse outcome for each item).
Change of stool type | 3 months
  Change of stool type evaluated by BRISTOL Stool Scale (range 1-7, lower and higher values representing worse outcome, middle values representing better outcome).
Change of serum concentration of IS and pCS | 3 months
  Change of free and total indoxyl sulfate (IS) and p-cresyl sulfate (pCS) serum concentrations (μg/mL) assessed by liquid chromatography/mass spectrometry
Change of serum concentration of inflammatory markers | 3 months
  Change of serum concentrations of interleukins: IL-6, TNF-α, IL-1, IL-8, IL-10 (pg/mL) evaluated by ELISA
Change of blood glucose level | 3 months
  Change of glycemia concentration (mg/dl)
Change of insulin levels | 3 months
  Change of insulin concentration (pmol/L)
Change of endocrine parameters | 3 months
  Change of C-peptide, growth hormone (GH), insulin-like growth factor 1 (IGF-1), testosterone concentration (ng/mL)
Change of serum concentration of D-lactate | 3 months
  Change of D-lactate serum concentration (uM)

OTHER OUTCOMES:
Gut microbiota | 3 months
  Change of the relative abundance (%) of Operational Taxonomic Units (OTUs) of Firmicutes, Bacteroidetes,Proteobacteria, Verrucomicrobia, Actinobacteria, Synergistetes, Cyanobacteria, Euryarchaeota, Chloroflexi, Nitrospirae, Tenericutes, Fusobacteria, Thermotogae, Acidobacteria evaluated by fecal bacterial DNA genome sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Loreto Gesualdo, MD Full Prof, Principal Investigator — Nephrology, Dialysis and Transplantation Unit "Aldo Moro" University of Bari
Locations (1):
- AOUConsorziale Policlinico Di Bari, Bari, Italy